CLINICAL TRIAL: NCT05089422
Title: Study of Clinical Types and Surgical Out Come of Pediatic Exotropia
Brief Title: Study of Clinical Types and Surgical Out Come of Pediatric Exotropia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sara Ali Hashim, ophthalmology resident doctor , principal investigator, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SAHashim
Record Dates: First submitted 2021-09-05; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Exotropia
MeSH Terms: conditions — Exotropia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with exotropia (Experimental): squint surgery
  Interventions: Procedure: Squint surgery

INTERVENTIONS:
Procedure: Squint surgery — Lateral rectus recession and /or medial rectus resection

SUMMARY:
study aiming to evaluate all children presented to strabismus clinic in ophthalmology department at sohag university hospital with divergent squint (exotropia) and to record surgical outcome of those who underwent strabismus surgery in our hospital

DETAILED DESCRIPTION:
A hospital-based, prospective, interventional study include infants and children up to the age of 15 years with Primary Concomitant divergent squint (1ry concomitant exotropia),Candidate for surgical correction of squint.

Each patient will be subjected to Detailed history and Full preoperative ophthalmic & orthoptic evaluation including: Visual acuity , ocular motility in the 6 cardinal directions, Hirschberg test & angle of deviation.

,Cover test & prism cover test for distant & near fixation,Cycloplegic refraction , Anterior segment examination, fundus examination.

_ post operative Follow-up regimen:

1. Children will be examined after surgery on: 1st postoperative day, 1st week, 1st month, 3rd month, and 6 months postoperatively.
2. The following will be recorded for each patient: Visual acuity, cover test, ocular motility testing, cover test and prism cover test, the degree of postoperative eye position, presence of over-correction or under-correction, and presence of any other complications.

ELIGIBILITY:
Inclusion Criteria:

1. Infants and children up to the age of 15 years.
2. Primary Concomitant divergent squint (1ry concomitant exotropia)
3. Candidate for surgical correction of squint

Exclusion Criteria:

1. Children with:

   1. Paralytic squint
   2. Consecutive exotropia
   3. Any neurological disorder
   4. History of previous squint surgery
   5. History of previous other ocular surgery (e.g. congenital cataract & glaucoma)
2. Children who missed follow up.

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
The number of children who become corrected post operatively | Six months
  Results of exotropia surgeries in children in sohag university hospital
The number of children with post operative residual squint | Six months
  Results of exotropia surgeries in children in sohag university hospital